CLINICAL TRIAL: NCT04757779
Title: A Single-arm, Phase Ⅱ Clinical Trial of Anlotinib Hydrochloride Combined With Irinotecan or Docetaxel for Second Line Treatment of Nonsensitive Relapsed Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZCH-2019-004
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Relapsed Small Cell Lung Cancer; Anlotinib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Docetaxel

STUDY DESIGN:
Intervention Model Description: From the start of the study, the subjects are orally administered with anlotinib 12mg on empty stomach. Subjects need to take anlotinib 2 weeks continuously and stop for 1 week(every 3 weeks is a cycle). On Day1 and Day8, subjects are required to inject irinotecan (65mg/m2) or docetaxel(60mg/m2) of a cycle,until disease progression or intolerable toxicity, for 4 cycles at most.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anlotinib hydrochloride combined with irinotecan or docetaxel (Experimental): From the start of the study, the subjects are orally administered with anlotinib 12mg on empty stomach. Subjects need to take anlotinib 2 weeks continuously and stop for 1 week(every 3 weeks is a cycle). On Day1 and Day8, subjects are required to inject irinotecan(65mg/m2) or docetaxel(60mg/m2) of a cycle,until disease progression or intolerable toxicity, for 4 cycles at most.
  Interventions: Drug: anlotinib hydrochloride combined with irinotecan or docetaxel

INTERVENTIONS:
Drug: anlotinib hydrochloride combined with irinotecan or docetaxel — From the start of the study, the subjects are orally administered with anlotinib 12mg on empty stomach.Subjects need to take anlotinib 2 weeks continuously and stop for 1 week(every 3 weeks is a cycle),the dose of anlotinib can be adjusted as 12mg,10mg or 8mg according to adverse effects.On Day1 and Day8, subjects are required to inject irinotecan (65mg/m2)or docetaxel (60mg/m2) of a cycle,until disease progression or intolerable toxicity, for 4 cycles at most.

SUMMARY:
Anlotinib hydrochloride is a multi-target antiangiogenic drug. It was recommended by Chinese Society of Clinical Oncology(CSCO) guideline as a third-line treatment for advanced small-cell lung cancer. This study intends to assess the efficacy and safety of anlotinib hydrochloride combined with irinotecan or docetaxel for second line treatment of nonsensitive relapsed small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject volunteered to participate in the study with informed consent signed.
2. Histologically or pathologically confirmed small-cell lung cancer (whether limited or advanced stage).
3. Have received at least first-line platinum-based chemotherapy for small-cell lung cancer and comfirmed disease relapse with imaging material. Disease progression during previous chemotherapy or less than 6 month after last chemotherapy.
4. Relapsed advanced small-cell lung cancer patients with symptom-controlled brain metastasis or leptomeningeal metastasis (subjects with symptomatic brain metastasis are allowed to receive radiotherapy, whether brain lesions can be deemed as target lesions is decided by investigators.); or patients with newly- discovered brain metastasis or leptomeningeal metastasis diagnosed by CT/MRI. Symptomatic or asymptomatic serosal cavity effusion (pleural effusion, ascites, pericardial effusion, local therapy is allowed). Radiotherapy for symptomatic bone metastasis or elsewhere is allowed as long as response evaluation is not affected.
5. Age:18-75 years old.
6. Eastern Cooperative Oncology Group (ECOG) performance status(PS) score ≤ 2.
7. Survival is expected to be ≥ 6 months.
8. At least one non-irradiated target lesion confirmed by CT/MRI scan less than 28 days before first dose of the study drug.
9. Male and women must use contraception within first dose to 24 weeks after last dose.
10. Major organ functions meet the following criteria within 7 days prior to treatment: blood routine examination and coagulation function (no blood transfusion within 14 days): hemoglobin≥90g/L; Absolute Neutrophil Count(ANC)≥1.5×109/L; Platelet (PLT)≥80×109/L; International normalized ratio(INR)≤1.5，Activated partial thromboplastin time(APTT)≤1.5 × upper limit of normal value(ULN); biochemical test standards: Total bilirubin(TBIL)≤1.5× ULN; ALT/AST≤2.5×ULN without liver metastasis, ALT/AST≤5×ULN with liver metastasis; Creatinine ≤1.25× ULN or endogenous creatinine clearance rate(Ccr)>45ml/min.

Exclusion Criteria:

1. Non-small-cell lung cancer (including a mixture of small-cell and non-small cell lung cancer).
2. Patients with small-cell lung cancer who relapsed more than 6 months after first- line treatment.
3. Medical imaging shows that the distance between the tumor and large vessels is less than 5mm; or lesions invade major blood vessels; or patients who are at risk of severe bleeding during the following treatment which is determined by investigators.
4. Medical imaging shows significant pulmonary cavity or necrotic tumor.
5. Uncontrolled hypertension (systolic blood pressure≥140mmHg or diastolic blood pressure≥90mmHg, even with optimal medication treatment).
6. Subjects with ≥grade Ⅱmyocardial ischemia or myocardial infarction, uncontrolled arrhythmia (include QT interval≥450ms for males, ≥470ms for females).
7. Heart function of NYHA grade Ⅲ-Ⅳ or left ventricle ejection fraction(LVEF)<50% confirmed by echocardiography.
8. Coagulant function abnormality (INR>1.5 or PT>ULN+4 seconds or APTT> 1.5ULN), with a bleeding tendency or patients is receiving thrombolytic or anticoagulant therapy.
9. For subjects who are using an anticoagulant or vitamin K antagonist (e.g. warfarin or heparin or other similar drugs), low dose heparin (6000-12000U daily for an adult) or aspirin (≤100mg daily) is allowed for preventive purposes when INR≤1.5.
10. Symptoms or propensity to bleed within 3 months prior to screening (include gastrointestinal hemorrhage, ulcerative gastric bleeding, fecal occult blood 2+ or above, vasculitis).
11. Arterial/venous thrombosis within 12 months prior to screening, e.g. cerebrovascular accident (include temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, pulmonary embolism.
12. Inherited or acquired bleeding and thrombus propensity (hemophilia, coagulation dysfunction, thrombocytopenia and hypersplenism).
13. Unhealed wound or fracture for a long time.
14. Major surgical operation or severe traumatic injury, bone fracture or ulcer within 4 weeks prior to screening, which affect drug absorption e.g. inability to swallow, chronic diarrhea and intestinal obstruction.
15. Abdominal fistula, gastrointestinal perforation, intraperitoneal abscess within 6 months prior to screening; routine urine test indicate urine protein≥++ or 24- hours proteinuria≥1.0g.
16. History of psychotropic drug abuse and cannot abstain from it or with mental disorders.
17. Participation in other clinical trials of anti-tumor drugs within 4 weeks prior to screening.
18. Previous or concurrent with other types of uncured malignancies, with the exception of cured basal cell carcinoma of the skin, carcinoma in situ of cervix and superficial bladder cancer.
19. Pregnant or lactating women, fertile patients who are unwilling or unable to use effective contraceptives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | 2 years
  the proportion of patients assessed with complete response and partial response

SECONDARY OUTCOMES:
progression-free survival time（PFS） | 2 years
  the time from date of randomization to disease progression or death
disease control rate（DCR） | 2 years
  the proportion of patients assessed with complete response，partial response and stable disease
overall survival（OS） | 2 years
  the time from date of randomization to death from any cause
quality of life（QoF）assessed by EORTC QLQ-C30 | 2 years
  Quality of Life assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30(EORTC QLQ-C30)
quality of life（QoF）assessed by EORTC QLQ LC-13 | 2 years
  Quality of Life assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer (EORTC QLQ LC-13)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hangzhou Cancer Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Tang Y, Liang J, Zhu L, Wang B, Pan K, Xu X, Chen X, Xia B. Combination of anlotinib and irinotecan as second-line therapy in extensive-stage small-cell lung cancer relapsed within six months: a single-arm phase Ⅱ study. Lung Cancer. 2025 Jul;205:108630. doi: 10.1016/j.lungcan.2025.108630. Epub 2025 Jun 20. PMID 40555062